CLINICAL TRIAL: NCT04553510
Title: Treatment of Bevacizumab Followed by Steroid in Radiation-induceded Brain Injury：a Randomized，Controlled and Single-blind Clinical Trail
Brief Title: Treatment of Bevacizumab Followed by Steroid in RN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160101; SYS-2016004 (Registry Identifier: Sun Yat-sen Memorial Hospital, Neurology department)
Record Dates: First submitted 2017-05-05; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Carcinoma; Adverse Effect of Radiation Therapy; Brain Injuries
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Radiation Injuries; Brain Injuries | interventions — Bevacizumab; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab and steroid (Experimental): Bevacizumab 5mg / kg, once every two weeks, a total of 6 weeks of 4 courses, sequential prednisone 10mg / d orally, the total course of 12 weeks.
  Interventions: Drug: Bevacizumab and steroid
- Bevacizumab and placebo (Active Comparator): Bevacizumab 5mg / kg, once every two weeks, a total of 6 weeks of 4 courses, sequential placebo 2 pills per day orally, the total course of 12 weeks.
  Interventions: Drug: Bevacizumab and placebo

INTERVENTIONS:
Drug: Bevacizumab and steroid — Bevacizumab 5mg / kg, once every two weeks, a total of 6 weeks of 4 courses, sequential prednisone 10mg / d orally, the total course of 12 weeks.
  Arms: Bevacizumab and steroid
Drug: Bevacizumab and placebo — Bevacizumab 5mg / kg, once every two weeks, a total of 6 weeks of 4 courses, sequential placebo 2 pills per day orally, the total course of 12 weeks.
  Arms: Bevacizumab and placebo

SUMMARY:
Treatment of bevacizumab followed by steroid may have a better effect on patients with radiation-induced brain injury.This randomized trial aims to investigate whether treatment of bevacizumab followed by steroid may alleviate radiation-induced brain injury in patients with nasopharyngeal carcinoma. The effect will be compared with outcomes in patients receiving steroid therapy

DETAILED DESCRIPTION:
Radiation-induced brain injury is a severe complication of radiotherapy in patients with Nasopharyngeal carcinoma. Current neuroprotective therapies show limited benefit in ameliorating this complication of radiotherapy. This study is a randomized, single blind clinical study. The primary aim of this study is to determine whether treatment of bevacizumab followed by steroid can alleviate radiation-induced brain injury in patients with nasopharyngeal carcinoma, and to compare the treating effect between combination of bevacizumab and steroid and bevacizumab alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received radiotherapy for histologically confirmed nasopharyngeal carcinoma.
2. Prior irradiation >/= 6 months prior to study entry.
3. Radiographic evidence to support the diagnosis of radiation-induced brain necrosis without tumor recurrence.
4. Age>/= 18 years. Because on dosing or adverse event data are currently not available on the use of bevacizumab in patients <18years old.
5. No prior bevacizumab therapy.
6. No evidence of very high intracranial pressure that suggests brain hernia and needs surgery.
7. Fertile women who are willing to take contraception during the trial.
8. Routine laboratory studies with bilirubin </=2 * upper limits of normal (ULN), aspartate aminotransferase (AST or SGOT) < 2 * ULN, creatinine <1.5 * ULN, red-cell count >/= 4,000 per cubic millimeter; white-cell count >/=1500 per cubic millimeter, platelets >/= 75,000 per cubic millimeter; Hb >/=9.0. PT, APTT, INR in a normal range.
9. If with history of seizures, patients should be on anticonvulsant therapy. However, preference will be enzyme-non-inducing anticonvulsants.
10. Ability to understand and willingness to sign a written informed consent document.
11. The patient has no active bleeding or pathological condition that carries a high risk of bleeding; there is no evidence of serious or non-healing wound, ulcer or bone fracture.

Exclusion Criteria:

1. evidence of metastatic disease;
2. evidence of tumor invasion to major vessels(e.g. the carotid);
3. history of bleeding related to tumor or radiotherapy during or after the completion of radiation.
4. Evidence of active central nervous system hemorrhage.
5. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to study enrollment.
6. inadequately controlled hypertension (systolic blood pressure (SBP) > 140 mmHg and/or diastolic blood pressure (DBP) > 90 mmHg despite antihypertensive medication)
7. Severe complications: 1) History of large vessel cerebrovascular accident (CVA) within 6 months; 2) Myocardial infarction or unstable angina within 6 months; 3) New York heart association grade II or greater congestive heart failure; 4) Serious and inadequately controlled cardiac arrhythmia; 5) Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection); 6) Clinically significant peripheral vascular disease; 7) severe infection.
8. Evidence of bleeding diathesis or coagulopathy.
9. Patients who have received steroid therapy for radiation-induced brain necrosis before the study.
10. History of anaphylactic response to bevacizumab.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in magnetic resonance imaging (MRI) of radiation-induced brain necrosis in patients | Change form baseline to evaluation at 12 weeks
  Change in MRI of radiation-induced brain necrosis in patients

SECONDARY OUTCOMES:
Change of neurologic function of patients after treatment | Change from baseline to evaluation at 12 weks.
  Change of neurologic function assessed using LENT/SOMA sacle of patients after treatment
Change of quality of life of patients after treatment | Change from baseline to evaluation at 12 weeks.
  Change of quality of life using QOL scale of patients after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tang Yamei, Ph.D, Study Director — sun yat-sen memorial hospital,sun yat-sen universicy
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No